CLINICAL TRIAL: NCT05573464
Title: A Randomized, Double-Blind, 12-Week (With an Extension to 52 Weeks in a Subset of Participants), Multi-Center Study to Assess the Safety of Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) Delivered by MDI HFO Compared to BGF Delivered by MDI HFA in Participants With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Assess the Safety of Budesonide/Glycopyrronium/Formoterol Fumarate With a Next-Generation Propellant in Participants With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5985C00003; 2022-001476-33 (EudraCT Number)
Record Dates: First submitted 2022-09-19; First posted 2022-10-10 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BGF MDI HFO 320/14.4/9.6μg (Experimental): Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) Delivered by MDI HFO (HFO-1234ze)
  Interventions: Drug: BGF MDI HFO 320/14.4/9.6 μg
- BGF MDI HFA 320/14.4/9.6 μg (Active Comparator): Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) Delivered by MDI HFA
  Interventions: Drug: BGF MDI HFA 320/14.4/9.6 μg

INTERVENTIONS:
Drug: BGF MDI HFO 320/14.4/9.6 μg — Budesonide, Glycopyrronium, and Formoterol Fumarate
  Other Names: BGF MDI HFO
  Arms: BGF MDI HFO 320/14.4/9.6μg
Drug: BGF MDI HFA 320/14.4/9.6 μg — Budesonide, Glycopyrronium, and Formoterol Fumarate
  Other Names: BGF MDI HFA
  Arms: BGF MDI HFA 320/14.4/9.6 μg

SUMMARY:
This is a 12-week (with an extension to 52 weeks in a subset of participants) study comparing the safety of BGF MDI HFO twice daily (BID) with BGF MDI HFA BID in participants with moderate to very severe COPD.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind, 12-week (with an extension to 52 weeks in a subset of participants) study comparing the safety of BGF MDI HFO 320/14.4/9.6 μg twice daily (BID) with BGF MDI HFA 320/14.4/9.6 μg BID in participants with moderate to very severe COPD. For the 12-week study, 542 participants will be randomized to treatments BGF MDI HFO and BGF MDI HFA in a 1:1 ratio. Randomization will be stratified by region (Americas, Europe) and COPD disease severity (percent predicted FEV1 ≥ 50%, percent predicted FEV1 < 50%). Subsequently, the 120 participants per treatment arm who were randomized to the extended study will continue and remain on the randomized treatment to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 40 to 80 years of age inclusive, at the time of signing the ICF;
2. Participants who have a documented history of physician-diagnosed COPD as defined by the ATS/ERS (Celli et al 2004) or by locally applicable guidelines;
3. Participants who have been regularly using dual ICS/LABA, LAMA/LABA, or ICS/LAMA/LABA (open or fixed-dose combinations) inhaled maintenance therapies for the management of their COPD for at least 6 weeks prior to Screening;
4. Participants who have pre-bronchodilator FEV1 of < 80% predicted normal at Visit 1;
5. Participants who have post-bronchodilator FEV1/FVC ratio of < 0.70 and post-bronchodilator FEV1 of ≥ 25% to < 80% predicted normal at Visit 2;
6. Participants who have CAT score ≥ 10 at Visit 1;
7. Participants who are current/former smokers with a history of at least 10 pack-years of tobacco smoking (1 pack year = 20 cigarettes smoked per day for 1 year);
8. Participants who are willing and, in the opinion of the Investigator, able to adjust current COPD therapy, as required by the protocol;
9. Participants must be able to demonstrate acceptable MDI administration and spirometry technique;
10. Participants who are willing to remain at the study center as required per protocol to complete all visit assessments;
11. Females must either be not of childbearing potential, or using a form of highly effective birth control as defined below:

    * Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:
    * Women < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) or more following cessation of exogenous hormonal treatment and follicle stimulating hormone levels in the postmenopausal range.
    * Women ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 52 weeks (12 months) or more following cessation of all exogenous hormonal treatment.
12. Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. At enrollment, women of childbearing potential who are sexually active with a non-sterilized male partner should be stable on their chosen method of highly effective birth control, as defined below, and willing to remain on the birth control until at least 14 days after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.

    * All women of childbearing potential must have a negative serum pregnancy test result at Visit 1
    * Women <50 years of age with amenorrhea for 12 months without an alternative medical cause must have a serum LH and FSH test (within 21-28 days before Visit 3) for study eligibility

    Highly effective birth control methods are listed below:
    * Sexual abstinence defined as complete abstinence from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant
    * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
    * Oral
    * Intravaginal
    * Transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation:
    * Oral
    * Injectable
    * Implantable
    * Intrauterine device or intrauterine hormone-releasing system
    * Male partner sterilization/vasectomy with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis or medical history interview provided by her or her partner.
    * Bilateral tubal ligation
13. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol

Exclusion Criteria:

1. Participants who have a documented history of physician-diagnosed asthma in the opinion of the Investigator based on thorough review of medical history and medical records, within 5 years of Visit 1;
2. Participants who have COPD due to α1-Antitrypsin Deficiency;
3. Participants with historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neurological, endocrine, gastrointestinal, or pulmonary. Significant is defined as any uncontrolled disease or any disease that, in the opinion of the Investigator, would put the safety of the participant at risk through participation, or that could affect the efficacy or safety analyses;
4. Sleep apnea that, in the opinion of the Investigator, cannot be controlled;
5. Other respiratory disorders including known active tuberculosis, lung cancer, cystic fibrosis, significant bronchiectasis (high resolution CT evidence of bronchiectasis that causes repeated acute exacerbations), immune deficiency disorders, severe neurological disorders affecting control of the upper airway, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or pulmonary thromboembolic disease;
6. Participant with moderate or severe COPD exacerbation or respiratory infection ending within 4 weeks prior to Visit 1 or during the Screening period;
7. Participant who has had a SARS-CoV-2 infection in the 8 weeks prior to Visit 1 or during the Screening Period or that required hospitalization at any time prior to Visit 1 or during the Screening Period;
8. Pulmonary resection or lung volume reduction surgery during the 26 weeks (6 months) prior to Visit 1 (ie, lobectomy, bronchoscopy lung volume reduction [endobronchial blockers, airway bypass, endobronchial valves, thermal vapor ablation, biological sealants, and airway implants]);
9. Long-term oxygen therapy;
10. Imminent life-threatening COPD (eg, need for mechanical ventilation);
11. Participant who has significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the Investigator, or any other relevant cardiovascular disorder as judged by the Investigator;
12. Participant with narrow angle glaucoma not adequately treated and/or change in vision that may be relevant, in the opinion of the Investigator; Note: All medications approved for control of intraocular pressures are allowed including topical ophthalmic nonselective beta-blockers and prostaglandin analogs.
13. Symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that, in the opinion of the Investigator, is clinically significant; Note: Participants with trans-urethral resection of prostate or full resection of the prostate within 26 weeks (6 months) prior to Visit 1 are excluded from the study
14. Unresectable cancer that has not been in complete remission for at least 5 years prior to Visit 1; Note: Squamous cell and basal cell carcinomas of the skin are not exclusionary
15. Known history of drug or alcohol abuse within 52 weeks (12 months) of Visit 1;
16. Unable to withhold short-acting bronchodilators for 6 hours prior to lung function testing at each applicable study visit;
17. Participant is unable to abstain from protocol-defined prohibited medications during Screening and Treatment Periods;
18. Using any herbal products either by inhalation or nebulizer within 2 weeks of Visit 1 and does not agree to stop for the duration of the study;
19. Participants with a known hypersensitivity to beta2-agonists, muscarinic antagonists, or corticosteroids, or any component of the MDI;
20. Participation in another clinical study with an intervention administered in the last 30 days or 5 half-lives, whichever is longer;
21. Previous randomization in any study using BGF MDI HFO (budesonide/glycopyrronium/formoterol fumarate - HFO);
22. Participants with calculated eGFR ≤ 30 mL/minute/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula;
23. Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, vital signs, or ECG, which in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study; Note: Participants with ECG QTcF interval (corrected for heart rate using Fridericia's formula [QTcF]) > 480 msec will be excluded. Participants with high degree atrioventricular block II or III, or with sinus node dysfunction with clinically significant pauses who are not treated with pacemaker will also be excluded.
24. Planned hospitalization during the study;
25. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site);
26. Study Investigators, sub-Investigators, coordinators, and their employee or immediate family members;
27. Judgment by the Investigator that the participant is unlikely to comply with study procedures, restrictions and requirements;
28. For women only - currently pregnant (confirmed with positive pregnancy test), breast feeding, or planned pregnancy during the study or women of childbearing potential not using acceptable contraception measures (see Inclusion criterion 12 in Section 5.1).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 559 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (20):
  - Research Site, Phoenix, Arizona
  - Research Site, Newport Beach, California
  - Research Site, Miami, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Valparaiso, Indiana
  - Research Site, Crowley, Louisiana
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Charlotte, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Dublin, Ohio
  - Research Site, Grants Pass, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Gaffney, South Carolina
  - Research Site, Longview, Texas
  - Research Site, McKinney, Texas
  - Research Site, Richmond, Virginia
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Fernando
- Bulgaria (9):
  - Research Site, Blagoevgrad
  - Research Site, Dupnitsa
  - Research Site, Lom
  - Research Site, Pernik
  - Research Site, Sandanski
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
  - Research Site, Vidin
- Canada (8):
  - Research Site, Truro, Nova Scotia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Germany (14):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Elsterwerda
  - Research Site, Essen
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Karlsruhe
  - Research Site, Koblenz
  - Research Site, Magdeburg
  - Research Site, Rheine
  - Research Site, Schwerin
  - Research Site, Wiesbaden
  - Research Site, Witten
- Mexico (5):
  - Research Site, Cuernavaca
  - Research Site, Culiacán
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
- Poland (12):
  - Research Site, Będzin
  - Research Site, Bydgoszcz
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Inowrocław
  - Research Site, Jelenia Góra
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Piaseczno
  - Research Site, Skórzewo
  - Research Site, Szczecin
  - Research Site, Zamość
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Mersin
  - Research Site, Pamukkale
- United Kingdom (5):
  - Research Site, Blackpool
  - Research Site, Corby
  - Research Site, Liverpool
  - Research Site, Poole
  - Research Site, Thetford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Usmani OS, Martinez FJ, Pandya H, Camiolo M, Bednarczyk A, Kucz K, Kokot M, Gottfridsson C, Aurivillius M, Pettersson L, Mei J, Skansen K, Bell JL, Petullo D, Collison K, Bondarov P, Jassal M, Patel M. Safety of budesonide/glycopyrronium/formoterol fumarate dihydrate delivered by HFO-1234ze versus HFA-134a in chronic obstructive pulmonary disease: a phase 3, multi-site, randomised, double-blind, parallel-group, active-comparator study. EClinicalMedicine. 2025 Aug 12;87:103402. doi: 10.1016/j.eclinm.2025.103402. eCollection 2025 Sep. PMID 40831469
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00003&attachmentIdentifier=e9beddc3-5afd-4d54-adec-6f1e29f41a25&fileName=CSR_Synopsis_.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants randomized were enrolled in the 12-week study. Of these, 120 participants in each arm were assigned (on first-in-study basis) to continue in the extended 52-week study. This is why the number who Started the 52-week treatment period is less than the Protocol Enrollment number.
Groups:
- BGF MDI HFO 320/14.4/9.6 μg: Budesonide, Glycopyrronium, and Formoterol Fumarate (BGF) Delivered by MDI HFO (HFO-1234ze)
Period: 12-week Treatment Period
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Started (Subjects randomised) | 280 | 279
Started Treatment | 280 | 278
Completed (Subjects who completed the 12-week treatment period) | 235 | 257
Not Completed | 45 | 22
Not completed — Discontinued intervention - other reason | 10 | 4
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Protocol Violation | 3 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 20 | 9
Not completed — Protocol-specified withdrawal criterion met | 1 | 0
Not completed — Randomised, not treated | 0 | 1
Period: 52-week Treatment Period
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Started (Assigned 52 weeks of treatment) | 120 | 120
Assigned 52 Weeks of Treatment and Started Treatment | 120 | 120
Completed (Completed 52 weeks of treatment) | 86 | 94
Not Completed | 34 | 26
Not completed — Discontinued intervention - other reason | 9 | 8
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 11 | 8
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Population: Overall number is based on the 12-week safety analysis set. This is defined as all participants who were randomised to study treatment and received at least one inhalation of study drug, irrespective of their protocol adherence and whether they would continue treatment for a total of 52-weeks. Participants will be analysed according to their treatment received. The actual treatment is defined as the study treatment that the participant received the most.
Groups:
- Total: Total of all reporting groups
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg | Total
Number analyzed (Participants) | 280 | 278 | 558
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 91 | 177
  >=65 years | 194 | 187 | 381
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.7) | 67.0 (7.0) | 67.0 (7.4)
Age, Continuous [Median (Full Range); unit: years] | 68.5 [41 to 80] | 68.0 [45 to 80] | 68.0 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 131 | 243
  Male | 168 | 147 | 315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 49 | 92
  Not Hispanic or Latino | 237 | 228 | 465
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 273 | 272 | 545
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events
Description: To assess the safety and tolerability of BGF MDI HFO as compared to BGF MDI HFA in participants with moderate to very severe COPD
Time Frame: Over 12 weeks
Population: 12-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 280 | 278
Participants
  Any serious adverse event | 15 | 12
  No serious adverse events | 265 | 266

2. Primary Outcome: Number and Percentage of Participants With Serious Adverse Events
Description: as for outcome 1
Time Frame: Over 52 weeks
Population: 52-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 120 | 120
Participants
  Any serious adverse event | 17 | 16
  No serious adverse events | 103 | 104

3. Primary Outcome: Number and Percentage of Participants With Non-serious Adverse Events >5%
Description: as for outcome 1
Time Frame: Over 12 weeks
Population: 12-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 280 | 278
Participants
  Any non-serious adverse event at the threshold cut-off greater than 5% | 46 | 47
  No non-serious adverse events at the threshold cut-off greater than 5% | 234 | 231

4. Primary Outcome: Number and Percentage of Participants With Non-serious Adverse Events >5%
Description: as for outcome 1
Time Frame: Over 52 weeks
Population: 52-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 120 | 120
Participants
  Any non-serious adverse event at the threshold cut-off greater than 5% | 46 | 67
  No non-serious adverse events at the threshold cut-off greater than 5% | 74 | 53

5. Primary Outcome: Number and Percentage of Participants With Adverse Events of Special Interest
Description: To assess the safety and tolerability of BGF MDI HFO as compared to BGF MDI HFA in participants with moderate to very severe COPD. Adverse events of special interest in this study are respiratory events such as dysphonia, cough, dyspnea, wheezing, paradoxical bronchospasm, bronchospasm, and COPD exacerbations.
Time Frame: Over 12 weeks
Population: 12-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 280 | 278
Participants
  Any adverse event of special interest | 52 | 55
  No adverse events of special interest | 228 | 223

6. Primary Outcome: Number and Percentage of Participants With Adverse Events of Special Interest
Description: as for outcome 5
Time Frame: Over 52 weeks
Population: 52-week safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
Number analyzed (Participants) | 120 | 120
Participants
  Any adverse event of special interest | 40 | 47
  No adverse events of special interest | 80 | 73

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | BGF MDI HFO 320/14.4/9.6 μg | BGF MDI HFA 320/14.4/9.6 μg
All-Cause Mortality (participants affected / at risk) | 1/280 | 1/278
Serious Adverse Events (participants affected / at risk) | 25/280 | 24/278
Other Adverse Events (participants affected / at risk) | 64/280 | 80/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI HFO 320/14.4/9.6 μg (N=280) | BGF MDI HFA 320/14.4/9.6 μg (N=278)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Trigeminal palsy (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Vertebral lateral recess stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI HFO 320/14.4/9.6 μg (N=280) | BGF MDI HFA 320/14.4/9.6 μg (N=278)
Nasopharyngitis (Infections and infestations) | 20 (24) | 30 (39)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 52 (68) | 60 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may not independently publish results until one of the following occurs: 1. multicentre primary publication is published; 2. no multicentre primary publication is submitted within 2 years after conclusion; 3. Sponsor confirms in writing there will be no multicentre primary publication.

PI shall provide the Sponsor with copies of any materials relating to the study that they intend to publish or make presentations relating to, at least 30 days in advance.

DOCUMENTS (2):
  • Study Protocol (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT05573464/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT05573464/SAP_001.pdf